CLINICAL TRIAL: NCT07067216
Title: Combined Effect of Biofeedback and Scapular Stabilization Exercises in Children With Swimmer's Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Osama Ali Hamed Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004998
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Swimmer Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Designed scapular stabilization using pressure biofeedback (Experimental): This group will consist of 20 participants, who will receive a designed scapular stabilization exercise program using pressure biofeedback. The program will be applied for one hour, two times per week, for 6 successive weeks.
  Interventions: Other: Designed scapular stabilization using pressure biofeedback
- Designed physical therapy program (Active Comparator): This group will consist of 20 participants, who will receive a designed physical therapy program. The program will be applied for one hour, two times per week, for 6 successive weeks.
  Interventions: Other: Designed physical therapy program

INTERVENTIONS:
Other: Designed scapular stabilization using pressure biofeedback — Patients will attend 1-hour physical therapy sessions twice weekly for 6 weeks. The program will include posterior capsule mobilization, scapular stabilization using pressure biofeedback (targeting lower trapezius, latissimus dorsi, pectoralis major, deep cervical flexors, and scapular retractors), and strengthening exercises using therabands: external rotation, shoulder diagonals, rows, and extensions. Additional training will involve physioball scapular exercises (up/down & side/side), prone scapular strengthening (e.g., TYI, superman), and scapular-clock drills to improve mobility, proprioception, and stability.
  Arms: Designed scapular stabilization using pressure biofeedback
Other: Designed physical therapy program — Patients will receive cryotherapy and perform stretching exercises for the pectoralis minor and posterior capsule. Strengthening exercises using theraband will target the rotator cuff (especially external rotators) and scapular depressors/retractors. Scapular stabilization will be trained through prone exercises on a ball (T, Y, W) and on a plinth, including rowing, horizontal abduction, extension, superman, and TYI exercises. Additionally, patients will perform the scapular-clock exercise to enhance mobility, control, and proprioception.
  Arms: Designed physical therapy program

SUMMARY:
The purpose of this study is to investigate the combined effect of biofeedback and scapular stabilization exercises on swimmer's shoulder in pediatric elite swimmers.

DETAILED DESCRIPTION:
Swimmer's shoulder is the most common injury in swimmers and is defined as a painful syndrome that occurs mostly in the anterior region of the shoulder and results from repetitive impingement of the rotator cuff under the coracoacromial arch during the technical gesture of swimming.

Shoulder injuries have been reported in up to 90% of swimmers. The scapula is vital in shoulder function and abnormal scapulothoracic mechanics and scapula-humeral rhythm have been implicated in shoulder pathologies, including glenohumeral impingement and rotator cuff tears.

When weakness or dysfunction is present in the scapular musculature, normal scapular positioning and mechanics may become altered which result in abnormal stresses to the capsular structures, rotator cuff compression and reduced performance.

Knowledge of scapulothoracic movements is regarded as crucial in the development of preventative strategies and treatment programs in athletes with shoulder pathology.

Scapula upward rotation is the dominant scapula action throughout shoulder elevation and has been previously implicated in the development of impingement.

In swimming, an athlete's scapular musculature plays a pivotal role in stabilizing and preventing impingement because its continuous activation is required throughout the swim stroke.

During all movements of the glenohumeral joint especially overhead elevation of the arm, it is of great importance that the scapular- stabilizing musculature should be strong enough to properly position the scapula. The main scapula stabilizers are the Levator Scapulae, Rhomboids major and minor, Serratus anterior, and Trapezii. These muscle groups function through synergistic co- contraction with rotator cuff to control the scapular movement. Scapular stabilization exercise aims to restore scapular position, orientations, motor control of muscles, and movement pattern, thereby attaining stability of scapula for better kinematics of shoulder. Due to lack of research area of scapular stabilization using a pressure biofeedback on swimmer's shoulder in pediatric swimmers, so the purpose of the study is to investigate the combined effect of scapular stabilization and biofeedback in children with swimmer's shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes form 9-13 years old and active in competitive swimming clubs
* Swimming styles will be selected are butterfly and backstroke styles and the swimmers undergone an average minimum of 4 hours of swimming per week.
* All pediatric swimmers have shoulder pain.
* All of them are not allowed to practice swimming during study.

Exclusion Criteria:

* Pediatric swimmers who practice any sport related to overhead activities.
* Swimmers who had dermatological problems.
* Past history of upper limb fractures or surgeries.
* Swimmers who had any neurological condition (like winging scapula due to nerve damage).
* Swimmers who had dorsal scoliosis (s or c shaped).
* Swimmers who integrate in swimming competitions at the same time of study.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-12 (Estimated); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 6 weeks
  The SPADI uses a 10 cm visual analogue scale for each question, with anchors from "no pain/difficulty" to "worst pain imaginable/so difficult it required help." Pain (5 items) and disability (8 items) scores are calculated separately and converted to percentages: pain (/50), disability (/80), and total SPADI (/130). If questions are skipped, scores are divided by the total possible. The final score (0-100) reflects shoulder impairment, with higher scores indicating worse function. A change of at least 13 points is needed to be considered meaningful beyond measurement error.

SECONDARY OUTCOMES:
Digital Inclinometer | 6 weeks
  Scapular upward rotation will be assessed in the scapular plane at humeral elevation angles of 0°, 60°, 90°, and 120°. Humeral angles will be set using an inclinometer along the upper arm. Subjects will elevate their arm with the thumb up, using a wall as a guide, and hold each position while scapular rotation is measured using a digital level placed over the scapula. Measurements will follow a sequence (0°-120°), with one trial per angle. Locator rods will be placed on the posterolateral acromion and scapular spine root. Subjects will return to rest and take 20-60 seconds breaks between trials to avoid fatigue.
Digital goniometer | 6 weeks
  Isolated glenohumeral internal-external rotation and elevation range of motion will be measured using standard techniques. Subjects will lie supine with the humerus at 90° abduction, neutral rotation, and the elbow flexed at 90°. The examiner will passively move the arm into internal or external rotation until a clinical endpoint is reached, then record the angle using a goniometer. These measurements will reflect pure glenohumeral motion by stabilizing the scapula during the assessment.
Kibler's Test (Lateral Scapular Slide Test) | 6 weeks
  This test assesses scapular symmetry using a reference point on the nearest spinous process to the scapula's inferior angle. Measurements are taken with arms at rest, then with hands on hips (~45° abduction), and finally at 90° elevation with maximal internal rotation (thumb to floor). Each position increases muscular demand. Distances from the reference point to the inferior angles of both scapulae are compared. A difference ≥1 cm is clinically significant; 1.5 cm is considered abnormal, and up to 3 cm may be seen with pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Nanees Essam Mohamed Salem, PhD, Study Chair — Professor, Cairo university; Shimaa Mohamed Reffat, PhD, Study Director — Assistant Professor, Cairo university
Locations (1):
- EL Hawar and Geziret Elward sporting clubs, Al Mansurah, Egypt